CLINICAL TRIAL: NCT03201835
Title: A Single-Center, Randomized, 5-Way Crossover Study to Compare the Safety, Tolerability and Pharmacokinetics of New Oral Cannabinoid Formulations Administered as Single Doses, With Buccal Sativex®, in Healthy Volunteers
Brief Title: 5-Way Crossover Study to Compare the Safety, Tolerability and Pharmacokinetics of New Oral Cannabinoid Formulations Administered as Single Doses, With Buccal Sativex®, in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PhytoTech Therapeutics, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CS-PYL-001
Record Dates: First submitted 2017-06-13; First posted 2017-06-28 (Actual); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — nabiximols

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- PNL-THC:CBD soft gelatin capsule (Experimental): 3 soft capsules, containing a total of 10.8 mg THC and 10 mg CBD (Each capsule contains 3.6 mg THC and 3.3 mg CBD)
  Interventions: Drug: PNL-THC:CBD soft gelatin capsule
- P-PNL-THC:CBD soft gelatin capsule (Experimental): 2 soft capsules containing a total of 7.2 mg THC, 6.7 mg CBD and 20 mg piperine (Each capsule contains 3.6 mg THC, 3.3 mg CBD and 10 mg piperine)
  Interventions: Drug: P-PNL-THC:CBD soft gelatin capsule
- CBD hard capsule dose 1 (Experimental): 1 hard capsule containing 10 mg CBD
  Interventions: Drug: CBD hard capsule dose 1
- CBD hard capsule dose 2 (Experimental): 1 hard capsule containing 100 mg CBD
  Interventions: Drug: CBD hard capsule dose 2
- Sativex® (Active Comparator): spray X 4 actuations, Each 100 μL spray contains 2.7 mg THC and 2.5 mg CBD, total per administration: 10.8 mg THC and 10 mg CBD
  Interventions: Drug: Sativex

INTERVENTIONS:
Drug: PNL-THC:CBD soft gelatin capsule — 3 soft capsules, containing a total of 10.8 mg THC and 10 mg CBD (Each capsule contains 3.6 mg THC and 3.3 mg CBD)
  Arms: PNL-THC:CBD soft gelatin capsule
Drug: Sativex — spray X 4 actuations
  Arms: Sativex®
Drug: CBD hard capsule dose 1 — 1 hard capsule containing 10 mg CBD
  Arms: CBD hard capsule dose 1
Drug: P-PNL-THC:CBD soft gelatin capsule — 2 soft capsules containing a total of 7.2 mg THC, 6.7 mg CBD and 20 mg piperine (Each capsule contains 3.6 mg THC, 3.3 mg CBD and 10 mg piperine)
  Arms: P-PNL-THC:CBD soft gelatin capsule
Drug: CBD hard capsule dose 2 — 1 hard capsule containing 100 mg CBD
  Arms: CBD hard capsule dose 2

SUMMARY:
The primary objective of the study was to evaluate the safety and tolerability of novel oral capsules containing THC and/or CBD, following a single administration to healthy volunteers. The secondary objective of the study was to compare the pharmacokinetic profiles of THC, THC metabolite 11-hydroxy-THC and/or CBD following a single administration of the investigational oral formulations with Sativex® Oromucosal Spray.

DETAILED DESCRIPTION:
Fifteen (15) healthy male volunteers received, following an overnight fasting and a standard breakfast, a single dose of either one of five administrations: PNL-THC:CBD, P-PNL-THC:CBD, CBD10 hard capsule, CBD100 hard capsule, Sativex® spray X 4. There was a wash-out period of no less than 4 days between each dosing.

Subjects underwent screening procedures within 21 days prior to first dosing, to assess their eligibility to participate in the study. Eligible subjects were admitted to the Clinical Research Center (CRC) in the evening before each study drug administration and will remained in-house for 24 hours after dosing. Following an overnight fast of at least 10 hours, the subjects received a standard meal within 30 minutes prior to dosing. Blood samples for PK were drawn at the specified time points. The subjects were monitored for safety, and AEs were recorded throughout the study. An End-of Study (EOS)/Safety Follow-up visit took place on 7-10 days after the last dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men between 18 and 45 years (inclusive) of age.
2. Subjects who provide written informed consent to participate in the study.
3. Body Mass Index (BMI) 19 to <30 kg/m2 and weight ranging between 65-85 kg.
4. Non-smoking and no use of any tobacco or nicotine products (by declaration) for a period of at least 6 months prior to screening visit
5. Subjects in general good health in the opinion of the investigator as determined by medical history, vital signs and a physical examination.
6. Supine blood pressure and heart rate within normal limits (blood pressure: systolic 90-140 mmHg; diastolic 50-90 mmHg, heart rate 50- 100 beats per minute (bpm)) on Screening visit.
7. Electrocardiogram (ECG) with no clinically significant abnormalities recorded at screening visit. Investigator assessment/discretion in cases of borderline results is allowed.
8. Negative HIV, Hepatitis B and Hepatitis C serology tests at screening.
9. No clinically significant abnormalities in hematology, blood chemistry, or urinalysis lab tests at screening.
10. No known history of alcohol or drug abuse. Negative urinary screen for drugs of abuse determined on Screening visit and on admission before each dosing (urine THC will be measured only before first dosing).
11. Subjects must be able to understand the requirements of the study and must be willing to comply with the requirements of the study.
12. Subjects must agree to abstain from driving from first drug administration until 3 weeks after last dosing.
13. Subject must agree not to engage in potentially hazardous activities such as operating machinery, working at heights (e.g. maintenance and construction, climbing a ladder) throughout the study duration.
14. Willing to abstain from cannabis use 30 days before and throughout the study duration.

Exclusion Criteria:

1. Known hypersensitivity to cannabinoids (including cannabis extracts), excipients or capsules.
2. Any history of adverse events associated with cannabis intoxication or dependence.
3. Known/suspected history or family history of psychiatric disorders
4. History of fainting or recurrent dizziness
5. History of epilepsy/seizures.
6. Documented history or ongoing symptoms of any gastrointestinal disorder involving motility, gastric acid or gastric emptying or malabsorption, including but not limited to, peptic ulcer disease, gastroesophageal reflux, dyspepsia, gastroparesis, chronic diarrhea, chronic constipation, gall bladder disease, pancreatitis, lactose intolerance and celiac disease.
7. History of esophageal, gastric, biliary, or intestinal surgery (excluding herniotomy and appendectomy which are not related to gastrointestinal disorders).
8. Known history of significant medical disorder, which in the investigator's judgment contraindicates administration of the study medications.
9. Presence of mouth ulcerations or any abnormalities of the oral cavity.
10. Any clinically significant abnormality upon physical examination or in the clinical laboratory tests at screening visit.
11. Used cannabinoids or a cannabinoid-based medicine within 30 days prior to receiving study medication.
12. Use of any prescription or over-the-counter (OTC) medications, vitamins and herbal or dietary supplements within 14 days prior to anticipated first dosing; subjects who had treatment with any known enzyme-altering agent (e.g. CYP450 inducers or inhibitors), within 30 days of first dosing. Paracetamol or for symptomatic relief of pain is allowed until 24 hours prior to first study drug administration.
13. Known drug hypersensitivity or history of idiosyncratic reactions to any drug.
14. Subjects with an abnormal diet, who had made substantial changes to eating habits within 30 days of the study,
15. History of drug or alcohol abuse in the last two years.
16. Any acute illness (e.g. acute infection) within 48 hours prior to the first study drug administration that is considered of significance by the investigator.
17. Participation in another clinical trial with drugs received within 3 months prior to first dosing (calculated from the previous study's last dosing date).
18. Subjects who donated blood in the 3 months or received blood or plasma derivatives in the 6 months preceding study drug administration.
19. Subjects who refuse to avoid strenuous physical activity within 48 hours prior to each drug administration and throughout in-house stay in the CRC.
20. Subjects with an inability to communicate well with the investigators and CRC staff (i.e., language problem, poor mental development or impaired cerebral function).
21. Subjects who are non-cooperative or unwilling to sign informed consent form.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-09-24 (Actual); Primary Completion 2015-12-06 (Actual); Study Completion 2016-06-06 (Actual)

PRIMARY OUTCOMES:
Frequency, severity, and duration of adverse events (AEs), including clinically significant laboratory abnormalities after administration of the study drugs | during 8 weeks from screening
  To evaluate the safety and tolerability of novel oral capsules containing THC and/or CBD, following a single administration to healthy volunteers. By evaluating frequency, severity, and duration of adverse events (AEs), including clinically significant laboratory abnormalities after administration of the study drugs

SECONDARY OUTCOMES:
Calculating pharmacokinetics Tmax | 0-24 hours for each treatmet arm
  To compare the pharmacokinetic profiles of THC, THC metabolite 11-hydroxy-THC and/or CBD following a single administration of the investigational oral formulations with Sativex® Oromucosal Spray, The following parameters will be evaluated for each subject's plasma:Tmax.
Calculating pharmacokinetics Cmax | 0-24 hours for each treatmet arm
  To compare the pharmacokinetic profiles of THC, THC metabolite 11-hydroxy-THC and/or CBD following a single administration of the investigational oral formulations with Sativex® Oromucosal Spray, The following parameters will be evaluated for each subject's plasma: Cmax
Calculating pharmacokinetics AUCT | 0-24 hours for each treatmet arm
  To compare the pharmacokinetic profiles of THC, THC metabolite 11-hydroxy-THC and/or CBD following a single administration of the investigational oral formulations with Sativex® Oromucosal Spray, The following parameters will be evaluated for each subject's plasma: AUCT.
Calculating pharmacokinetics AUCInf | 0-24 hours for each treatmet arm
  To compare the pharmacokinetic profiles of THC, THC metabolite 11-hydroxy-THC and/or CBD following a single administration of the investigational oral formulations with Sativex® Oromucosal Spray, The following parameters will be evaluated for each subject's plasma: AUCInf
Calculating pharmacokinetics T½. | 0-24 hours for each treatmet arm
  To compare the pharmacokinetic profiles of THC, THC metabolite 11-hydroxy-THC and/or CBD following a single administration of the investigational oral formulations with Sativex® Oromucosal Spray, The following parameters will be evaluated for each subject's plasma: T½.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center (CRC)- Souraskey Medical center, Tel Aviv, Israel